CLINICAL TRIAL: NCT01290146
Title: Early Use of Levosimendan Compared to Usual Care in Advanced Chronic Heart Failure (ACHF)
Brief Title: ELEVATE Early LEvosimendan Vs Usual Care in Advanced Chronic hearT failurE
Acronym: ELEVATE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to lack of enrollment
Sponsor: Niguarda Hospital (Other)
Collaborators: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EudraCT code 2009-016958-41; FO002 (Registry Identifier: Ethics Committee)
Record Dates: First submitted 2011-02-03; First posted 2011-02-04 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Advanced Chronic Heart Failure
Keywords: Heart Failure; Levosimendan; Inotropic agents; Phosphodiesterase Inhibitors; Vasodilators; Diuretics
MeSH Terms: conditions — Heart Failure | interventions — Diuretics; Simendan

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diuretics (Active Comparator): Patients randomized to diuretics receive a 24-hour diuretic infusion with a maximum cumulative dose up to 200 mg furosemide/24 h
  Interventions: Drug: Diuretics
- Levosimendan (Experimental): Patients randomized to Levosimendan receive a 24-hour levosimendan infusion with NO prior bolus injection.
  Starting doses will be based on baseline SBP levels
  * SBP ≥ 85-99mmHg: 0.05 mcg/kg/min
  * SBP ≥100 mmHg: 0.1 mcg/kg/min
  Interventions: Drug: Levosimendan

INTERVENTIONS:
Drug: Diuretics — Patients randomized to diuretics receive a 24-hour diuretic infusion with a maximum cumulative dose up to 200 mg furosemide/24 h
  Arms: Diuretics
Drug: Levosimendan — Patients randomized to Levosimendan receive a 24-hour levosimendan infusion with NO prior bolus injection.
  Starting doses will be based on baseline SBP levels
  * SBP ≥ 85-99mmHg: 0.05 mcg/kg/min
  * SBP ≥100 mmHg: 0.1 mcg/kg/min
  Arms: Levosimendan

SUMMARY:
The purpose of this study is to compare in patients with Advanced Chronic Heart Failure the effects of Levosimendan versus diuretic (single 24-hour infusion) applied at the early detection of impending destabilization on hospitalization-free survival during 12 months.

Patients with advanced chronic heart failure (ACHF) have a short term reduced life expectancy with recurrent hospital admissions for clinical exacerbations. Levosimendan improves contractility by calcium-dependent binding to troponin C, determines vasodilation of the coronary arteries and systemic resistance vessels, thus decreasing preload and afterload, while exerting a protective effect on the myocardium against ischemia-reperfusion damage. In randomized clinical trials of acute heart failure patients, levosimendan improved hemodynamics and patients' quality of life and decreased natriuretic peptide plasma levels, with no excess mortality The study will assess whether the administration of levosimendan (single 24-hour infusion) at the early detection of deterioration may reduce frequency and duration of hospital admissions, improve functional status and quality of life in ACHF patients, with respect to diuretic infusion.

DETAILED DESCRIPTION:
BACKGROUND Patients with advanced chronic heart failure (ACHF) have a short term reduced life expectancy with recurrent hospital admissions for clinical exacerbations. ACHF poses a heavy burden to cardiology departments, where these patients are referred for the severity of their clinical condition, which require a specialist approach, and results in high health care costs due to frequent rehospitalizations.

Patients with ACHF ≥ 2 hospital admissions in 6 months are at high risk of recurrent exacerbations. The benefits of strict outpatient follow-up at specialised HF vs standard community care in ACHF patients have been consistently demonstrated. The standard approach at HF clinics is based on flexible diuretic dose and outpatient iv diuretics as bolus or infusion at early signs of decompensation. Although this strategy results in symptomatic benefit and prevents approximately one third of hospital admission for acute exacerbations, a relevant proportion of patients will still need hospitalization. Predictors of lack of benefit are low systolic blood pressure, prior increase in oral diuretics and beta-blocker use, which taken together represent markers of severe disease susceptible to evolve in a low output state.

In the HF clinic setting, a novel strategy for these patients, to include early support to myocardial contractility, i.e. before compelling criteria for hospital admission become manifest, might prevent further prolonged hospitalizations, myocardial damage and impairment in renal function TRIAL RATIONALE Levosimendan improved hemodynamics and patients' quality of life and decreased natriuretic peptide plasma levels, with no excess mortality, in randomized clinical trials of acute heart failure. In SURVIVE an early larger treatment effect of levosimendan was apparent in patients with acute worsening of chronic HF treatment than in those with de novo disease, possibly because a greater proportion of these patients may be on beta-blockers, that are known to interfere with dobutamine or may potentiate the circulatory actions of levosimendan. Thus levosimendan may be unattractive first-line agent in destabilized ACHF patients on beta-blockers.

Based on the drug cardioprotective properties, hemodynamic and neurohormonal effects, we propose a novel therapeutic approach for the clinically-driven use of levosimendan in recurrent acute exacerbations of ACHF.

Dosing of the drug will omit the bolus to increase tolerability in this severely ill patient population.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Systolic dysfunction (LVEF ≤ 35% by echo assessment within 6 months before enrolment)
* No requirement for hospital admission for diagnostic work up or elective treatment to define etiology and/or treatment plan
* Already on optimal standard HF treatment based on individual tolerance, including cardiac resynchronization therapy (CRT)/ICD device according to current guidelines
* At least 2 hospital admissions for HF in the 6 months before enrolment, the most recent one within 30-90 days before enrolment with requirement for inotrope administration

Exclusion Criteria:

* Participant in other studies in the last 30 days
* Life expectancy < 1 year for comorbid conditions other than HF
* Pregnancy, lactation, childbearing potential unless on adequate contraception
* Acute coronary syndromes, percutaneous or surgical revascularization, valve surgery performed within 8 weeks before enrolment
* Planned percutaneous or surgical procedures (except for heart transplantation)
* CRT within 6 months before enrolment
* Cardiogenic shock
* Supine systolic BP < 85 mmHg
* Severe liver insufficiency (>three-fold increase in AST-ALT )
* Sever chronic kidney dysfunction (estimated GFR < 30 ml/min)
* Sustained ventricular tachycardia
* Severe chronic or current acute infection (temperature >38 C, WBC >15,000/mm3)
* Severe chronic obstructive pulmonary disease (FEV1 <30% predicted or on oxygen therapy)
* Severe persistent anemia (Hb < 10 g/l))
* ACHF exacerbation due to conditions requiring specific treatment (e.g. anemia, atrial fibrillation, supraventricular tachycardia ) Documented low compliance or unavailable for programmed follow-up visits and phone contact

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2011-02 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Number of days alive free of Transplant and out-of-hospital (DAOH) | Measured at 12 months

SECONDARY OUTCOMES:
Incidence of acute renal dysfunction | Measured at at 24 hours since inception of randomized treatment for acute worsening HF
  proportion of subjects who develop AKIN stage 1 (increase > 0.3 mg/dl or > 25% in serum creatinine from previous visit)
All cause mortality, hospital readmission and unscheduled office and emergency department visits for ADCHF | Measured at 12 months
  A combination of all cause hospital admissions/death/urgent heart transplantation/LV assist device implantation
BNP changes | Measured at at end-of- study and at each eventual destabilization
  Percent changes in BNP vs baseline
Number of hospital admissions for acute worsening HF | Measured at 12 months
  Number of hospital admissions for acute worsening HF
Costs | Measured at 12 months
  Direct health care costs for days in hospital, supplementary visits, drug treatment
Treatment-related adverse events | Measured at 12 months
  death, hospital a dimission, emergency room or clinic unscheduled visits
Adverse changes in blood pressure or heart rate | Measured at 24 hours after iv treatment
  Hypotension (< 90 mmHg), tachycardia (> 110 bpm)
ECG changes | Measured at 24 hours after iv treatment
  Rhythm, rate, conduction disturbances, ventricular arrhythmias, repolarization changes

CONTACTS AND LOCATIONS:
Overall Officials: Fabrizio Oliva, MD, Study Chair — Heart Failure Heart Transplant Program, Cardiovascular Department, Niguarda Hospital, Milan, Italy; Michele Senni, MD, Study Chair — Cardiovascular Medicine Ospedali Riuniti, Bergamo, Italy
Locations (22):
- Italy (22):
  - Ospedali Riuniti di Ancona Cardiology Presidio Lancisi, Ancona, Ancona
  - Azienda Ospedaliero-Universitaria, Consorziale Policlinico di Bari, U.O. Cardiologia Universitaria, Dipartimento Emergenza e Trapianti di Organi, Bari, Bari
  - Fondazione S. Maugeri. IRCCS Istituto di Cassano Murge, Cassano Murge, Bari
  - Ospedali Riuniti di Bergamo Cardiovascular Medicine, Bergamo, Bergamo
  - Ospedale Brotzu Cardiology, Cagliari, Cagliari
  - Ospedale Sant'Anna Cardiology, Como, Como
  - Ospedale SS Annunziata Cardiology, Cosenza, Cosenza
  - Istituti Ospitalieri di Cremona Cardiology, Cremona, Cremona
  - Ospedale Santa Maria Nuova Cardiology, Florence, Firenze
  - Ospedale Vito Fazzi, Lecce, Lecce
  - Istituto Auxologico Italiano - IRCCS Clinical Cardiology Cardiovascular Department, Milan, Milan
  - Azienda Ospedaliera Niguarda Heart Failure and Heart Transplant Program, Milan, Milan
  - Azienda Ospedaliera S. Gerardo Hear Failure and Cardiomyopathy Clinic, Monza, Monza
  - Gruppo Policlinico di Monza Clinical Cardiology and Heart Failure Unit Cardiology Department, Monza, Monza
  - Ospedale Santa Maria della Misericordia Cardiology, Perugia, Perugia
  - Ospedale Guglielmo da Saliceto Cardiology Department, Piacenza, Piacenza
  - Azienda Ospedaliera San Camillo-Forlanini, Cardiology, Heart Failure Clinic, Roma, Roma
  - Università di Roma Sapienza Dipartimento di Scienze Cardiovascolari e Respiratorie, Roma, Roma
  - Azienda Ospedaliera San Giovanni- Addolorata 1st Cardiology Unit, Roma, Roma
  - Ospedale Santo Spirito, Cardiology, Roma, Roma
  - Azienda Ospedaliero-Universitaria, Ospedale di Cattinara Cardiology, Trieste, Trieste
  - Ospedale di Circolo e Fondazione Macchi Cardiology, Varese, Varese